CLINICAL TRIAL: NCT07083986
Title: Immediate and Long-term Results of Carotid Endarterectomy and Stenting in the Acute Stage of Ischemic Stroke
Brief Title: Carotid Endarterectomy Versus Stenting in Patients With Acute Stage of Ischemic Stroke.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Pryamikov Aleksandr, MD, PhD (DMedSc [Russia]), Associate Professor, Pirogov Russian National Research Medical University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 25225062025
Record Dates: First submitted 2025-07-05; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Ischaemic Stroke; Carotid Endarterectomy; Carotid Stenting
MeSH Terms: conditions — Ischemic Stroke | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients in acute period of Ischaemic Stroke (Experimental)
  Interventions: Procedure: Carotid Artery Stent Placement; Procedure: carotid endarterectomy

INTERVENTIONS:
Procedure: Carotid Artery Stent Placement — Carotid Artery Stent Placement was performed according to the standard technique.
Procedure: carotid endarterectomy — Carotid endarterectomy with stenting was performed according to the standard technique. For the purpose of the greatest comparability in the volume of anesthesia, it was decided to use regional anesthesia in all cases, including adequate dynamic observation of neurological status.

SUMMARY:
The objective of this clinical trial is to compare immediate and long-term results of carotid endarterectomy and carotid stenting in acute period of ischemic stroke. Patients who presented with acute stage of ischemic stroke will be treated by carotid artery stenting in 50 cases and by carotid endarterectomy in 50 cases under regional anesthesia.

Patient inclusion criteria:

1. Ischemic stroke in the middle cerebral artery territory
2. Ipsilateral stenosis of the internal carotid artery more than 50%
3. Neurological deficit at the time of surgical treatment: the modified Rankin scale (mRs) score of 0-4 and the US National Institutes of Health (NIHSS) stroke scale score no more than 12
4. The size of the ischemia focus: no more than 1/3 in the territory of the middle cerebral artery brain supply
5. Terms of operation: from 1 to 28 days from the moment of ischemic stroke

The primary intra-hospital and/or 30-day study endpoints:

1. Perioperative ipsilateral ischemic stroke.
2. Any stroke: contralateral ischemic or any hemorrhagic stroke.
3. Myocardial infarction.
4. Hemorrhagic complications that required surgical revision of the operating wound or transfusion of blood components.
5. Surgical site infection
6. Death
7. Main adverse cardiovascular events (stroke + myocardial infarction + death).

ELIGIBILITY:
Inclusion Criteria:

* 1. Ischemic stroke in the middle cerebral artery territory 2. Ipsilateral stenosis of the internal carotid artery more than 50% 3. Neurological deficit at the time of surgical treatment: the modified Rankin scale (mRs) score of 0-4 and the US National Institutes of Health (NIHSS) stroke scale score no more than 12 4. The size of the ischemia focus: no more than 1/3 in the territory of the middle cerebral artery brain supply 5. Terms of operation: from 1 to 28 days from the moment of ischemic strok

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2026-05-21 (Estimated); Study Completion 2028-05-21 (Estimated)

PRIMARY OUTCOMES:
Rate of Hemorrhagic complications (%) | "Baseline" "Perioperative/Periprocedural" "up to 30 day" "1 year" "through study completion, an average of 1 year".
  The primary outcome measure was 30-day postoperative intracerebral hemorrhage (ICH)
Rate of perioperative ipsilateral ischemic stroke (%) | "Baseline" "Perioperative/Periprocedural" "up to 30 day" "1 year" "through study completion, an average of 1 year".
  The primary endpoint was ipsilateral stroke < 30 days.
Rate of any stroke (%) | "Baseline" "Perioperative/Periprocedural" "up to 30 day" "1 year" "through study completion, an average of 1 year".
Rate of Myocardial infarction (%) | "Baseline" "Perioperative/Periprocedural" "up to 30 day" "1 year" "through study completion, an average of 1 year".
Rate of Surgical site infection (%) | "Baseline" "Perioperative/Periprocedural" "up to 30 day" "1 year" "through study completion, an average of 1 year".
Rate of Death (%) | "Baseline" "Perioperative/Periprocedural" "up to 30 day" "1 year" "through study completion, an average of 1 year".
Rate of main adverse cardiovascular events (%) | "Baseline" "Perioperative/Periprocedural" "up to 30 day" "1 year" "through study completion, an average of 1 year".

CONTACTS AND LOCATIONS:
Locations (1):
- Moscow City Clinical Hospital named after V.M. Buyanov, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes